CLINICAL TRIAL: NCT00891904
Title: A Feasibility Study of Re-irradiation Using Stereotactic Body Radiation Therapy (SBRT) and Cetuximab for Recurrent Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Radiation Therapy and Cetuximab in Treating Patients With Recurrent Head and Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000640992; RPCI-I-143108
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Results first posted 2014-03-12 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab (Experimental): Patients receive cetuximab IV over 60-120 minutes once weekly in weeks 1-5
  Interventions: Biological: cetuximab; Radiation: stereotactic body radiation therapy

INTERVENTIONS:
Biological: cetuximab — Given IV
Radiation: stereotactic body radiation therapy — Undergoing Radiotherapy

SUMMARY:
RATIONALE: Stereotactic body radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving stereotactic body radiation therapy together with cetuximab may kill more tumor cells.

PURPOSE: This clinical trial is studying the side effects of radiation therapy given together with cetuximab and to see how well it works in treating patients with recurrent head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the toxicity of stereotactic body radiotherapy delivered concurrently with cetuximab in patients with recurrent squamous cell carcinoma of the head and neck.

Secondary

* To assess the feasibility of delivering this regimen in these patients.
* To assess the impact of this regimen on local control, distant control, and overall survival of these patients.

OUTLINE: Patients receive cetuximab IV over 60-120 minutes once weekly in weeks 1-5. Patients undergo 1 fraction of stereotactic-body radiotherapy (RT) in week 2. At 4 weeks after RT completion, patients may receive additional cetuximab IV combined with a 28-day chemotherapy regimen, per investigator discretion.

After completion of study treatment, patients are followed every 2 months for 1 year, every 3-4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the oral cavity, paranasal sinuses, nasopharynx, larynx, hypopharynx, or oropharynx

  * Medically or surgically inoperable disease or patient refuses surgery
  * Recurrent disease
* Previously irradiated disease meeting the following criteria:

  * Prior radiotherapy completed > 6 months from re-irradiation
  * Prior radiotherapy in the region of the study cancer that would result in overlap of radiation therapy fields
  * Majority of the recurrent tumor volume (> 50%) received prior radiotherapy dose of 30-75 Gy
* No distant metastatic disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 60 days after completion of study treatment
* No prior allergic reaction to study drugs

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior surgical resection of the recurrent primary tumor and/or regional lymphatics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-04; Primary Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anurag K. Singh, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Biological/Vaccine: Cetuximab: All patients enrolled will receive cetuximab 400 mg/m 2 IV x 1 dose 1 week prior to delivery of SBRT. Patients will then receive 15 Gy x 1 using SBRT and cetuximab i.v.
  250 mg/m2 weekly for 4 weeks (total of 5 doses at 250 mg/m2).
Period: Overall Study
Arm/Group | Biological/Vaccine: Cetuximab
Started | 2
Completed | 0
Not Completed | 2
Not completed — Death | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Biological/Vaccine: Cetuximab
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (2.8)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Grade 4-5 Toxicity as Assessed by NCI CTCAE v.30
Time Frame: Daily while on Treatment
Population: Trial terminated early. Too few patients to analyze.
Arm/Group | Biological/Vaccine: Cetuximab
Number analyzed (Participants) | 0

2. Secondary Outcome: Feasibility as Assessed According to Ability to Deliver the Entire Treatment Regimen to 80% of Patients
Time Frame: 2 years
Population: Trial terminated early. Too few patients to analyze.
Arm/Group | Biological/Vaccine: Cetuximab
Number analyzed (Participants) | 0

3. Secondary Outcome: Local and Distant Control
Time Frame: very 2 months for year one, every 3-4 months for year 2, every 6 months for years 3 and 4 and annually thereafter.
Population: Trial terminated early. Too few patients to analyze.
Arm/Group | Biological/Vaccine: Cetuximab
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Time Frame: very 2 months for year one, every 3-4 months for year 2, every 6 months for years 3 and 4 and annually thereafter
Population: Trial terminated early. Too few patients to analyze.
Arm/Group | Biological/Vaccine: Cetuximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Biological/Vaccine: Cetuximab
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biological/Vaccine: Cetuximab (N=2)
Pneumonia (Infections and infestations) | 1 (2)
Postoperative wound infection (Infections and infestations) | 1 (4)
Alanine aminotransferase increased (Investigations) | 1 (4)
Aspartate aminotransferase increased (Investigations) | 1 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biological/Vaccine: Cetuximab (N=2)
White blood cell disorder (Blood and lymphatic system disorders) | 1 (4)
Nausea (Gastrointestinal disorders) | 1 (4)
Alanine aminotransferase increased (Investigations) | 1 (4)
Aspartate aminotransferase increased (Investigations) | 1 (4)
Haemoglobin decreased (Investigations) | 1 (4)
Neutrophil count decreased (Investigations) | 1 (8)
Platelet count decreased (Investigations) | 1 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (4)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (4)

LIMITATIONS AND CAVEATS:
Trial terminated early. Too few patients to analyze.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes